CLINICAL TRIAL: NCT06013475
Title: Use of Darolutamide, Enzalutamide and Apalutamide for Non-metastatic Castration-Resistant Prostate Cancer (nmCRPC) - EXTension of the DEAR Real-world Study (NCT05362149)
Brief Title: An Observational Cohort Study to Describe and Compare the Use of Darolutamide, Enzalutamide and Apalutamide and How Well These Work in Men With Non-metastatic Castration-resistant Prostate Cancer (nmCRPC) in Real World Settings
Acronym: DEAR-EXT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22625
Record Dates: First submitted 2023-08-18; First posted 2023-08-28 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Non-metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — apalutamide; darolutamide; enzalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Apalutamide
  Interventions: Drug: Apalutamide
- Darolutamide
  Interventions: Drug: Darolutamide (BAY 1841788)
- Enzalutamide
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Apalutamide — Decision by the treating physician
  Groups: Apalutamide
Drug: Darolutamide (BAY 1841788) — Decision by the treating physician
  Other Names: Nubeqa
  Groups: Darolutamide
Drug: Enzalutamide — Decision by treating physician
  Groups: Enzalutamide

SUMMARY:
This is an observational cohort study in men with non-metastatic castration-resistant prostate cancer who received their usual treatment, which is 'Androgen receptor inhibitors' (ARIs) including darolutamide, enzalutamide, and apalutamide.

The main purpose of this study is to collect data on the length of time men with nmCRPC continued treatment with darolutamide, enzalutamide, or apalutamide as prescribed by their doctors. Researchers will only include men who had not been treated with any new type of medication that blocks the action of hormones.

The data will come from an electronic health record database called Precision Point Specialty (PPS) Prostate Cancer Electronic Medical Record (EMR) for men in the United States of America. EMR data will be verified and supplemented via patient chart review. Data collected will be from January 2019 to September 2023. .

ELIGIBILITY:
Inclusion Criteria:

1. Men diagnosed with prostate cancer.
2. Diagnosis of nmCRPC prior to or within 90 days after the first ARI treatment initiation
3. Treatment with Darolutamide, Enzalutamide, or Apalutamide initiated for the first time
4. Age ≥ 18 years at treatment start
5. At least 6 months of Electro-Medical-Record activity after the treatment start unless the patient died earlier than 6 months.

Exclusion Criteria:

1. Evidence of metastatic disease before or 30 days after treatment start
2. Prior history of other primary cancers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men previously not treated with a novel antihormonal agent and starting the initial ARI treatment for nmCRPC during the study period, in US community urology practices
Sampling Method: Non-Probability Sample
Enrollment: 1375 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Time to ARI treatment discontinuation | Retrospective analysis from 01-Aug-2019 to 30 Sep 2023

SECONDARY OUTCOMES:
Reasons for ARI treatment discontinuation | Retrospective analysis from 01-Aug-2019 to 30 Sep 2023
Proportion of patients, who switched to another ARI therapy | Retrospective analysis from 01-Aug-2019 to 30 Sep 2023
Frequency of adverse events | Retrospective analysis from 01-Aug-2019 to 30 Sep 2023
Time to progression to mCRPC | Retrospective analysis from 01-Aug-2019 to 30 Sep 2023
Dose modification of initial ARI | Retrospective analysis from 01-Aug-2019 to 30 Sep 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.